CLINICAL TRIAL: NCT00616252
Title: Comparison of the Pharmacokinetics of Antiretroviral Agents in HIV Infected Ugandan Women During and After Pregnancy
Brief Title: Antiretroviral Drug Levels During and After Pregnancy
Status: Completed | Type: Observational
Sponsor: Makerere University (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Dr Concepta Merry, Infectious Diseases Institute
Other Study IDs: CPR 002
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2010-12

CONDITIONS: Pharmacokinetics
Keywords: Antiretroviral; Pharmacokinetics; Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Human plasma Red cell pellets
Oversight: Data Monitoring Committee: No

SUMMARY:
In HIV-infected women, the use of combination therapy with antiretrovirals (ARV) in pregnancy prevents HIV related morbidity and mortality and prevents mother-to-child transmission of the HIV virus.

Specifically, suppression of the virus to an undetectable level is important during the delivery of the baby to minimize potential HIV exposure. In Sub-Saharan Africa, the use of ARV combinations containing nevirapine is the cornerstone of current HIV therapy, due to an affordable cost, availability in a fixed dose combination pill, and generic availability. Maintaining the efficacy and preventing development of resistance against this agent by the HIV virus is imperative, as second line therapies are often more difficult to obtain, are more expensive, and present more challenges in drug storage in clinics and in the community.

Pregnancy adds another dimension to the challenge of treating women with HIV, as the physiologic and metabolic changes can affect levels of antiretroviral agents in the body. Though these changes are known to exist, few trials have evaluated the effect of these factors on the pharmacokinetics of antiretroviral agents and their impact has yet to be demonstrated.

We wish to evaluate if the physiologic changes that occur during pregnancy impact the levels of stavudine, lamivudine, and nevirapine compared to those of a non-pregnant, HIV-infected Ugandan female. These data are imperative to ensure adequate suppression of the HIV virus throughout pregnancy.

DETAILED DESCRIPTION:
In HIV-infected women, the use of combination therapy with antiretrovirals (ARV) in pregnancy prevents HIV related morbidity and mortality and prevents mother-to-child transmission of the HIV virus.1 Specifically, suppression of the virus to an undetectable level is important during the delivery of the baby to minimize potential HIV exposure. Commonly prescribed ARV therapy in Ugandan pregnant women includes a combination of two NRTIs, along with a non-nucleoside reverse transcriptase inhibitor (NNRTI), nevirapine. In Sub-Saharan Africa, the use of nevirapine containing regimens is the cornerstone of current ARV therapy, due to an affordable cost, availability in a fixed dose combination pill, and generic availability. Maintaining the efficacy and preventing development of resistance against this agent by the HIV virus is imperative, as second line therapies are often more difficult to obtain, are more expensive, and present more challenges in drug storage in clinics and in the community.

Data have demonstrated that higher exposure to nevirapine is associated with a greater likelihood of achieving virologic control as well as maintaining virologic response over the long term, while sub-optimal drug levels may result in the development of viral resistance.2 The use of combination therapy is important due to the development of resistance seen using single dose therapy with nevirapine at delivery.3 Resistance to nevirapine is particularly worrisome due to the cross-resistance between nevirapine and other NNRTIs, potentially eliminating one essential class of ARVs used to treat HIV. Evaluating nevirapine exposure is also important to avoid toxicities related to excess levels of nevirapine, which may compromise patient adherence to the regimen and put the woman at risk for virologic failure in addition to increased drug toxicity.4, 5

To our knowledge, most studies to date have only evaluated the pharmacokinetics of first dose nevirapine in HIV-infected pregnant women during delivery.6,7 Other studies have had too few sampling times to fully characterize the pharmacokinetic parameters of nevirapine. However, previous studies have demonstrated that pharmacokinetic changes do occur with other ARVs metabolized by a metabolic path similar to nevirapine. For example, one published study demonstrated lower levels of nelfinavir and a disproportionate amount of the nelfinavir M8 metabolite in pregnant women during their third trimester, possibly implicating alterations in the cytochrome P450 enzyme system responsible for both nelfinavir and nevirapine metabolism.8, 9 Given this evidence with similarly metabolized drugs, it is important to definitively characterize nevirapine pharmacokinetics to ensure the safe use of this drug during pregnancy.

Data have also demonstrated a direct correlation between zidovudine intracellular triphosphate concentrations and change in CD4 cell count during therapy as well as a direct correlation between lamivudine intracellular triphosphate concentrations and decline in HIV RNA in plasma.10 Data have also shown that there is a wide inter-patient variability in the concentration of the NRTIs, and adjusting these concentrations based on therapeutic drug monitoring has resulted in improved virologic outcomes for patients.11, 12 No information is known about the intracellular triphosphorylated concentrations of the NRTIs in the pregnant female. We seek to establish if there is a necessity for further evaluation of intracellular levels of all NRTI agents in the pregnant population through this research.

The available pharmacokinetic data to date, have primarily evaluated male populations in the western world. We are just beginning to understand the complex pharmacogenomic mechanisms that play a role in pharmacokinetics and pharmacodynamics. Efavirenz, also an NNRTI, and nevirapine have both been identified as having different pharmacokinetic properties in African patients as compared to American, European, and South American patients.13,14 These changes will play a significant role in the long term efficacy and toxicity of these agents as they are used on a more widespread basis in Sub-Saharan Africa. Evaluating these changes in African women during pregnancy is also essential as females represent the predominant gender impacted by HIV in Sub-Saharan Africa. These changes during pregnancy may impact the safety of these agents in pregnant females if the levels are higher than expected, and may also impact the mother-to-child transmission rate and long term use of these agents if the levels are lower than desired.

Pregnancy adds another dimension to the challenge of treating women with HIV, as the physiologic and metabolic changes can impact the pharmacokinetics of antiretroviral agents. Proposed mechanisms include absorption changes due to prolonged gastric and intestinal emptying time, decreased gastric acid secretion, and increased mucus secretion; increased volume of distribution of drug caused by increased total body water and fat, and decreased plasma protein concentration; changes in elimination related to stimulation of hepatic microsomal enzymes and inhibition of microsomal oxidases; the effects of the fetus including compartmentalization of drugs in the fetus and placenta, biotransformation of drugs by the fetus and placenta, and additional elimination of drugs by the fetus.15,16 Though these physiologic and metabolic changes are known to exist, few trials have evaluated the effect of these factors on the pharmacokinetics of antiretroviral agents and their impact has yet to be demonstrated.

Few pharmacokinetic studies have been undertaken to date in Sub-Saharan Africa, though it is becoming recognized that in order to support the antiretroviral rollout program, these studies are essential for the safe and effective long-term use of these agents. The University of Makerere, Infectious Diseases Institute, is establishing a strong foundation for pharmacokinetic work to take place in Uganda through the development of a pharmacokinetic laboratory which will become the leading resource for pharmacokinetic work in Sub-Saharan Africa. This makes the Makerere University the logical location for this essential evaluation. One of the first studies evaluating pharmacokinetic parameters in African patients was performed by our co-investigators at the Joint Clinical Research Center in Kampala, and established that pharmacokinetic evaluation of these drugs in an African population is both necessary and logistically feasible(22) .

We wish to evaluate if the physiologic changes that occur during pregnancy impact the pharmacokinetics of stavudine, lamivudine, and nevirapine compared to those of a non-pregnant, HIV-infected Ugandan female. Evaluation of drug concentrations at steady state, instead of after a single dose is essential, as most patients are maintained on these medications throughout their pregnancy to ensure complete virologic suppression at the time of delivery. These data are imperative to ensure adequate viral suppression throughout pregnancy and to minimize the likelihood of the development of viral resistance engendered by inadequate drug concentrations

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected pregnant female in her second or third trimester who requires ARV therapy during her pregnancy
* Antiretroviral therapy includes nevirapine in addition to two NRTI agents
* Informed consent obtained

Exclusion Criteria:

* If primary physician feels the required blood draws would be potentially dangerous to the patient or fetus
* Haemoglobin <8 g/dL
* Liver Function tests > 2x normal
* CD4 cell count >250 cells/mL if ART naive
* Calculated Creatinine Clearance < 30 ml/min at any visit during the study period
* Patients receiving any medications that may interact with the cytochrome p450 enzyme system metabolism of nevirapine
* Concurrent herbal medication use.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: HIV positive women attending ante-natal care clinic at Mulago Hospital, Kampala Uganda
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2008-02; Primary Completion 2008-11 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To evaluate differences in the trough concentration (C12hr) of nevirapine during the second and third trimester of pregnancy and after delivery in the same patient | 12 months

SECONDARY OUTCOMES:
To evaluate differences in the clearance (Cl/F), area under the curve (AUC), Volume of distribution (V/F), maximum concentration (Cmax), time to maximum concentration (Tmax), and half-life (T1/2) of nevirapine as a result of pregnancy. | 12 months
To evaluate potential changes in intracellular triphosphate concentration of NRTIs that may occur as a result of pregnancy | 12 months
To evaluate pharmacogenomic differences in this East African population. | 12 months
To establish pharmacokinetic levels seen in non-pregnant East African women as compared to the levels seen in the western population, based on the post-partum levels. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Concepta A Merry, PhD, Principal Investigator — University of Dublin, Trinity College
Locations (1):
- Infectious Diseases Institute, Faculty of Medicine, Makerere University, Kampala, Kampala, Uganda